CLINICAL TRIAL: NCT07376980
Title: Modified Single-Stapled Anastomosis in Laparoscopic or Robotic Low Anterior Resection for Rectal Cancer: The SMART Trial (Single-Modified Anastomosis for Rectal Cancer Surgery Technique), A Multicenter Randomized Controlled Study
Brief Title: The SMART Trial: Modified Single-Stapled Anastomosis in Laparoscopic or Robotic Low Anterior Resection for Rectal Cancer
Acronym: MST
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Kyunghee University Medical Center (Other); Seoul National University Hospital (Other); Kyungpook National University Chilgok Hospital (Other); Saint Vincent's Hospital, Korea (Other); Sinchon Severance Hospital, Yonsei University College of Medicine (Unknown)
Responsible Party: Principal Investigator, Kim, Jin, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025AN0114
Record Dates: First submitted 2025-12-03; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Rectal Neoplasms; Rectal Neoplasms Malignant; Rectal Cancer; Rectal Cancer Surgery
Keywords: Rectal Cancer; Total Mesorectal Excision; Low Anterior Resection; Anastomotic Leak; Anastomosis, Surgical; Stapled anastomosis; Modified Single-Stapled Technique; Minimally Invasive Rectal Surgery
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment interventional model. Participants will be randomly allocated in a 1:1 ratio to one of two dependent surgical intervention arms: MST or DST. Each participatns will undergo only assigned surgical technique without crossover betwen groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: No additional parties.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified single-stapled anastomosis technique (Experimental): Participants assigned to this arm will undergo minimally invasive low anterior resection using the modified single-stapled technique. After rectal resection, the two ends of the linear staple line of stump are approximated toward the center using a barbed suture. The circular stapler spike is introduced through the center of the staple line to ensure complete resection of the linear staple line, eliminating staple-line intersections. The reaminder of the procedure, including total mesorectal excision, follows standard oncologic principles.
  Interventions: Procedure: Modified single-stapled anastomosis technique
- Double-stapled anastomosis technique (No Intervention): Participants assigned to this arm will undergo minimally invasive low anterior resection using the conventional double-stapled technique. The rectum is transected with linear stapler, followed by transanal introduction of a circular stapler to create an end-to-end anastomosis. The procedure represents current standard practice for low anterior resection in rectal cancer.

INTERVENTIONS:
Procedure: Modified single-stapled anastomosis technique — This intervention applies a modified single-stapled anastomosis specifically to low anterior resection (LAR), where the technique has not been previously evaluated in a randomized controlled trial. Although similar concepts have been explored in anterior resection, their application in LAR is technically more challenging due to the deeper pelvic working space and more limited access to the rectal stump. In earlier studies, approximation of the linear staple line was performed through a Pfannelstein incision or mini-laparotomy incision during specimen extraction. In contrast, this trial utilizes a fully intracorporeal approach.
  Other Names: Single-stapled anastomosis; Modified single-stapled anastomosis; Dog-ear-free anastomosis; Single-stapling technique; Modified double-stapling technique; Dog-ear closure technique
  Arms: Modified single-stapled anastomosis technique

SUMMARY:
The goal of this clinical trial is to learn whether a modified single-stapled anastomosis (MST) can reduce anastomotic leakage compared with the conventional double-stapled technique (DST) in adult patients undergoing laparoscopic or robotic low anterior resection for rectal cancer.

The main questions it aims to answer are:

* Does MST lower the incidence of anastomotic leakage after rectal cancer surgery?
* Does MST improve short-term surgical outcomes compared with DST?

Researchers will compare the MST group with the DST group to see if MST leads to fewer anastomotic leaks and safer postoperative recovery.

Participants will:

Receive either MST or DST during minimally invasive rectal cancer surgery Undergo routine postoperative CT scans within one month after surgery to check for symptomatic or asymptomatic anastomotic leakage Attend scheduled follow-up visits and standard postoperative assessments as part of routine rectal cancer care

DETAILED DESCRIPTION:
Anastomotic leakage is one of the most serious complications after low anterior resection (LAR) for rectal cancer. This complication can lead to infection, reoperation, prolonged hospitalization, higher medical costs, and worse long-term oncologic outcomes. Although laparoscopic and robotic surgery have improved short-term recovery compared with open surgery, the risk of anastomotic leakage remains a major concern.

The most commonly used reconstruction method during minimally invasive LAR is the double-stapled technique (DST). In DST, the rectum is transected with a linear stapler and then reconnected with a circular stapler. This creates an intersection between two staple lines, a known weak point that may be prone to leakage due to structural and ischemic vulnerability.

The modified single-stapled technique (MST) eliminates this intersection. Before applying the circular stapler, the two ends of the linear staple line on the rectal stump are brought together using a simple suture. This results in a single, centered staple line that the circular stapler incorporates completely into the anastomosis. Early studies, including a previous randomized trial, suggest that MST significantly reduces anastomotic leakage compared with DST.

This multicenter randomized controlled trial aims to provide high-quality evidence on the effectiveness of MST in reducing anastomotic leakage in patients undergoing laparoscopic or robotic LAR for rectal cancer. A total of 440 adult patients will be enrolled across multiple high-volume university hospitals in South Korea. Participants will be randomly assigned in a 1:1 ratio to receive MST or DST. Randomization will be stratified by sex, neoadjuvant treatment, and study center.

To ensure consistent surgical quality, all participating colorectal surgeons will complete a pre-trial standardization workshop and submit unedited surgical videos for competency review. All surgical procedures will follow standardized steps, and perioperative care will be based on established Enhanced Recovery After Surgery (ERAS) protocols.

The primary outcome is the rate of anastomotic leakage within one month after surgery. All participants will undergo routine abdominopelvic CT scans within this time window to detect both symptomatic and asymptomatic leaks. Secondary outcomes include postoperative complications, operative time, distal resection margin length, hospital stay, and long-term oncologic outcomes such as recurrence and survival. If MST is shown to be superior to DST, this study may support a simple, low-cost, and easily adoptable modification to current surgical practice. MST does not require additional equipment or complex training, making it a potentially valuable technique that can improve patient safety and surgical outcomes in rectal cancer care across diverse clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with rectal cancer who are scheduled to undergo laparoscopic or robotic low anterior resection
* histologically confirmed rectal adenocarcinoma located within 15cm from anal verge.
* ECOG performance status of 0 to 2
* Any clinical stage

Exclusion Criteria:

* Who have significant comorbidities or history of abdominal surgeries that would preclude a minimally invasive approach
* Bowel obstruction for perforation requiring emergency surgey
* Concurrent, or recent treatment for colorectal or other malignancies within the past five years
* Presence of inflammatory bowel diseases
* Hereditary colorectal cancer syndrome

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leakage | within 30 days after surgery
  Anastomotic leakage will be assessed within 30 days after surgery using clinical evaluation and routine abdominopelvic computed tomography (APCT). Leakage is defined as any defect in the anastomosis that results in communication between the inside of the bowel and the surrounding tissue. Diagnostic criteria include clinical symptoms (such as fever, abdominal pain, or drainage contents), abnormal laboratory findings, or radiologic evidence of leakage on APCT. All leaks will be classified according to the grading system.
  * Grade A: Leakage requiring no active therapeutic intervention.
  * Grade B: Leakage requiring non-surgical management, such as antibiotics or percutaneous drainage.
  * Grade C: Leakage requiring reoperation. Routine postoperative CT for all participants ensures consistent and standardized detection of both symptomatic and asymptomatic leaks.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Kim, M.D., Ph.D, Principal Investigator — Korea University Anam Hospital
Locations (6):
- South Korea (6):
  - St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Kyungpook National University Chilgok Hospital, Daegu, Gyeongsangbuk-do
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because the dataset contains sensitive clinical information, and secondary distribution is not permitted under the terms of institutional review board approvals and patient consent. Data access is restricted to the study investigators to protect participant privacy.